CLINICAL TRIAL: NCT02627664
Title: Prospective Study of Dysarthria, Swallowing Disorders and Respiratory in Parkinson's Disease
Brief Title: Study of Dysarthria, Swallowing Disorders and Respiratory in Parkinson's Disease
Acronym: ProdDiGYPark
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: France Parkinson Association (Other)
Responsible Party: Sponsor
Other Study IDs: 2010_21; 2010-A01391-38 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2014-12-18; First posted 2015-12-11 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Parkinson's Disease
Keywords: Idiopathic early; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observational study: natural history of non dopaminergic signs
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — natural history of non dopaminergic signs

SUMMARY:
The investigators prospectively enrolled 64 early PD patients (less than 3 years after the first symptom) in order to prospectively assess the natural history of non-dopaminergic symptoms.

DETAILED DESCRIPTION:
Patients were evaluated at baseline and after 2 years in off drug condition. Clinical, psychological, neuropsychological evaluations, functional respiratory evaluation, swallowing video fluoroscopy, dysarthria, gait and axial disorders.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic parkinson's disease

Exclusion Criteria:

* dementia
* severe axial gait disorders
* respiratory or ENT pathology
* Pregnancy

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease (PD) with early idiopathic ( ≤ 5 years of evolution )
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-02-09 (Actual)

PRIMARY OUTCOMES:
dysarthria severity assessed by the BECD scale | 2 years
  BECD (French battery of clinical evaluation of the dysarthria) is a validated scale for qualitative assessment of dysarthria severity in neurological disorders, especially PD

SECONDARY OUTCOMES:
respiratory insufficiency detection | 2 years
  pulmonary function tests include spirometry with standard spirometer and maximal inspiratory and expiratory flow volume curves . At least 3 reproductible F-V curves are necessary. Values of FCV, FEV, peak expiratory flow, peak inspiratory flow, forced expiratory flow, SNIP were measured 12 hours after last levodopa intake (off drug)
swallowing function | 2 years
  150 mL glass of water test video fluoroscopy of swallow in off drug condition face and profile incidences: qualitative analysis of oral, pharyngeal, aspiration if necessary blindly assessed by 2 ENT experts in PD
gait axial function (freezing) | 2 years
  SWS test rhythmic tests for differens imposed frequencies (upper lower limb and facial) kinematic analysis of gait parameters by VICON (oxford metrics)
Mattis scale | 2 years
LARS scale | 2 years
MADRS scale | 2 years
PAS scale | 2 years
MoCA | 2 years
Genetic Polymorphisme | 2 years
  To evaluate of cognitive and profile correlation to the polymorphisms of COMT (catechol-O-methyltransferase: Val158Met COMT) of MAPT H1 / H2 (microtubule associated tau protein) and ApoE (Apolipoprotein-E-ε2, 3, 4 )

CONTACTS AND LOCATIONS:
Overall Officials: luc defebvre, MD PhD, Study Chair — CHRU LILLE FRANCE
Locations (1):
- Francine Niset, Lille, France

IPD SHARING:
Plan to Share IPD: No